CLINICAL TRIAL: NCT00005889
Title: Study of Gluconeogenesis in Very Low Birth Weight Infants Receiving Total Parenteral Nutrition
Brief Title: Gluconeogenesis in Very Low Birth Weight Infants Who Are Receiving Nutrition By Intravenous Infusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00188-0667; BCM-H7213; BCM-GCRC-0667
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Infant, Low Birth Weight; Hyperglycemia
Keywords: endocrine disorders; hyperglycemia; low birth weight; neonatal disorders; rare disease
MeSH Terms: conditions — Hyperglycemia; Endocrine System Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Alanine; Amino Acids; Glucagon; Glucose; Glutamine; Glycerol; Insulin; Leucine; Lipids; Urea

INTERVENTIONS:
Drug: alanine
Drug: amino acids
Drug: glucagon
Drug: glucose
Drug: glutamine
Drug: glycerol
Drug: insulin
Drug: leucine
Drug: lipids
Drug: urea

SUMMARY:
RATIONALE: Very low birth weight infants have problems maintaining normal blood sugar levels. Gluconeogenesis is the production of sugar from amino acids and fats. The best combination of amino acids, fat, and sugar to help very low birth weigh infants maintain normal blood sugar levels is not yet known.

PURPOSE: Clinical trial to study how very low birth weight infants break down amino acids, fat, and sugar given by intravenous infusion, and the effect of different combinations of nutrients on the infants' ability to maintain normal blood sugar levels.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are assigned to one of 6 study groups.

Patients receive infusions of stable isotope tracers: [15N]urea IV beginning at -12 hours and continuing over 22 hours to measure protein oxidation; [U-13C]glucose IV beginning at zero hour and continuing over 10 hours to measure glucose appearance rate and gluconeogenesis; [2-13C]glycerol IV over 10 hours to measure lipolysis; and [1-C]leucine IV over 10 hours to measure proteolysis. Blood samples are obtained before the start of the urea tracer infusion; before the start of the glucose, glycerol, and leucine tracer infusions; and at study hours 4, 4.5, 5, 9, 9.5, and 10. Blood glucose is measured hourly, and patients receive glucose IV if blood glucose falls below 40 mg/dL.

Group I: Patients are randomized to one of two study arms. Arm I: Patients receive standard total parenteral nutrition (TPN), except the [U-13C]glucose is substituted for a portion of the glucose. Arm II: The infusions of lipids (Intralipid) and amino acids (TrophAmine) are discontinued at study hour zero. The infusion rate of natural glucose will be reduced during the first hour, and thereafter discontinued.

Group II: Patients are randomized to receive either TrophAmine or Intralipid IV over the last 5 hours of the study.

Group III: Patients are randomized to receive one of two different doses of glycerol IV over the last 5 hours of the study.

Group IV: Patients are randomized to receive either glutamine or alanine IV over the last 5 hours of the study.

Group V: Patients receive glucagon IV for 24 hours prior to study. Patients are then randomized to receive glucagon IV with either IV glucose alone or with Intralipid and TrophAmine IV.

Group VI: Patients who are hyperglycemic receive TPN and [U-13C]glucose as in group I, arm I, over 14 hours, and regular insulin IV at 10 hours, followed by an IV infusion of carbohydrate. Blood samples obtained between hours 4 and 5 are omitted, and are drawn instead between hours 13 and 14.

ELIGIBILITY:
* Clinically stable, very low birth weight infants (750-1,500 grams)
* Normal blood glucose values OR Blood glucose greater than 175 mg/dL
* No prior insulin
* No sepsis Oxygen supply less than 30% Normal acid base status
* No malformation
* No discernible diseases

Ages: 4 Days to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Agneta L. Sunehag, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765